CLINICAL TRIAL: NCT04293042
Title: A Pilot Study in the Treatment of BK Virus Infection With Cytotoxic T Cells in Immunocompromised Transplant Patients
Brief Title: Treatment of BK Virus Infection With CTL Cells in Immunocompromised Transplant Patients
Acronym: BK-CTLs
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Caitlin Elgarten, Attending Physician, Assistant Professor, Perelman School of Medicine at the University of Pennsylvania, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-016545
Record Dates: First submitted 2020-01-23; First posted 2020-03-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: BK Polyomavirus

STUDY DESIGN:
Intervention Model Description: This open-label, single-arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BK cystitis and/or nephropathy (Experimental): All patients with symptoms that are consistent with BK cystitis and/or nephropathy (frequency, dysuria, hematuria, elevated creatinine) will have serum quantitative DNA PCR for BK virus level measured in log copies per mL (results also expressed in copies per milliliter), performed in the Children's Hospital of Philadelphia Infectious Disease Diagnostics Laboratory
  Interventions: Biological: BK-virus specific CTLs

INTERVENTIONS:
Biological: BK-virus specific CTLs — HLA Matched Related Donors: BK-virus specific CTLs (2.5 x 104 CD3/kg) infused intravenously on day 0 and may be additionally reinfused at a minimum of every two weeks (depending on safety and efficacy) for a maximum of five total infusions (maximum 12.5 x 104 CD3/kg).
  HLA Mismatched Related Donors: BK-virus specific CTLs (0.5x104 CD3/kg) infused intravenously on day 0 and may additionally be reinfused at a minimum of every two weeks (depending on safety and efficacy) for a maximum of five total infusions (maximum 2.5 x 104 CD3/kg).

SUMMARY:
This is a pilot study using cytotoxic T lymphocytes (CTLs) manufactured with the Miltenyi CliniMACS Prodigy Gamma-capture system will be effective in decreasing specific viral load in patients with BK virus viremia and BK virus-associated symptoms post-allogeneic hematopoietic stem cell transplantation (HSCT), renal transplantation, and chemotherapy.

DETAILED DESCRIPTION:
This open-label, single-arm clinical trial will assess the safety and efficacy of BK virus-specific CTLs isolated from whole blood or leukapheresis products. The BK virus -specific CTLs will be generated automatically by the CliniMACS® Prodigy using the CliniMACS Cytokine Capture System (IFNgamma) after incubation with MACS GMP PepTivator® Peptide Pools of BKV VP1 and BKV LT.

ELIGIBILITY:
Inclusion Criteria:

Patient Eligibility

* Patients with symptoms of cystitis and elevated BK virus DNA by screening PCR as above (section 4) post allogeneic HSCT, post chemotherapy

  1. Symptoms of cystitis may include: hematuria (microscopic or gross), pain with urination, frequency, bladder spasms.
  2. Patient may be otherwise treated for cystitis as per local institutional standards. Such treatments may include hydration, antiviral medications, or surgical intervention as deemed appropriate by treating physician.
* Consent: Written informed consent given (by patient or legal representative) prior to any study-related procedures.
* Performance Status > 30% (Lansky < 16 yrs and Karnofsky > 16 yrs)
* Age: 0.1 to 25 years
* Females of childbearing potential with a negative urine pregnancy test.

Donor Eligibility

* Related donor available with a T-cell response to the BK-virus MACS® PepTivator® antigen(s).

  1. Original allogeneic donor if available, IgG positive for BKV or confirmatory testing to respond to BKV MACS Peptivator®.
  2. Third Party Allogeneic Donor: If original donor is not available or does not have a T-cell response: third party allogeneic donor (family donor > 1 HLA A, B, DR match to recipient) with a T-cell response to the BK MACS® PepTivator.

     AND
* Allogeneic donor disease screening is complete similar to hematopoietic stem cell donors (Appendix 1).

AND

• Obtained informed consents by donor or donor legally authorized representative prior to donor collection.

Exclusion Criteria:

Patient exclusion criteria:

A patient meeting any of the following criteria is not eligible for the present study:

* Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of BK Virus CTL infusion
* Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of BK Virus CTL infusion or within 3 days of planned infusion.
* Thymoglobulin (ATG), campath or T cell immunosuppressive monoclonal antibodies within 30 days
* Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30%
* Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory BK virus infection.
* Any medical condition which could compromise participation in the study according to the investigator's assessment
* Known HIV infection
* Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.
* Known hypersensitivity to iron dextran
* Patients unwilling or unable to comply with the protocol or unable to give informed consent.
* Known human anti-mouse antibodies

Ages: 5 Weeks to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Grade III-IV acute GVHD | Up to 8 weeks after last BK-CTL infusion
  Number of participants with Grade III-IV acute GVHD as assessed by CTCAE v4.0
Number of patients with undetectable BK viral load | 12 weeks after first BK-CTL infusion
  Number of patients with undetectable BK viral load as measured by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Elgarten, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No